CLINICAL TRIAL: NCT03203317
Title: Insulin-dependent and Exercise-induced Myocellular Signalling in Skeletal Muscle
Brief Title: Myocellular Signalling in Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Nielsen, Assistant Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TIN-X
Record Dates: First submitted 2017-04-26; First posted 2017-06-29 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Exercise; Insulin Sensitivity
MeSH Terms: conditions — Motor Activity; Insulin Resistance | interventions — Insulin; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin-stimulation (Experimental): 2 h insulin-clamp
  Interventions: Drug: Insulin
- Exercise (Experimental): 10 min of maximal exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Drug: Insulin — 2 h insulin clamp
  Arms: Insulin-stimulation
Other: Exercise — Cycling exercise
  Arms: Exercise

SUMMARY:
The study will investigate myocellular signalling in skeletal muscle after insulin-stimulation and exercise in healthy young men

ELIGIBILITY:
Inclusion Criteria:

* healthy
* informed consent
* habitual training (2-5 h/week)
* VO2max of 40-60 ml/min/kg
* lean mass 55-65 kg

Exclusion Criteria:

* smoker
* allergy towards insulin
* chronic disease

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Change in muscle phospho-proteome signature | Before and after 10 minutes of exercise, as well as before and after a 2 hour insulin stimulation
  proteomic analysis of mixed muscle homogenate

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenahgen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided